CLINICAL TRIAL: NCT04162210
Title: A Phase III, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of Single Agent Belantamab Mafodotin Compared to Pomalidomide Plus Lowdose Dexamethasone (Pom/Dex) in Participants With Relapsed/Refractory Multiple Myeloma (RRMM) (DREAMM 3)
Brief Title: Study of Single Agent Belantamab Mafodotin Versus Pomalidomide Plus Low-dose Dexamethasone (Pom/Dex) in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)
Acronym: DREAMM-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207495; 2018-004252-38 (EudraCT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Belantamab mafodotin; Pomalidomide; Dexamethasone; Relapsed/Refractory Multiple Myeloma; Driving Excellence in Approaches to Multiple Myeloma 3 (DREAMM 3)
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized and multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Belantamab mafodotin (Experimental): Participants will receive belantamab mafodotin single agent dose on Day 1 of Q3W
  Interventions: Drug: Belantamab mafodotin
- Participants receiving pom/dex (Active Comparator): Participants will receive pomalidomide daily on Days 1 to 21 of each 28-day cycle, with dexamethasone once weekly on Days 1, 8, 15 and 22.
  Interventions: Drug: Pom/dex (Pomalidomide plus low dose Dexamethasone)

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
  Arms: Participants receiving Belantamab mafodotin
Drug: Pom/dex (Pomalidomide plus low dose Dexamethasone) — Pomalidomide and Dexamethasone will be administered.
  Arms: Participants receiving pom/dex

SUMMARY:
This open-label, randomized study for evaluating the efficacy and safety of single agent belantamab mafodotin when compared to pom/dex in participants with RRMM. Participants will be randomized in a 2:1 ratio to receive either single agent belantamab mafodotin or pom/dex. Belantamab mafodotin will be administered on Day 1 (D1) at every 3 weeks (Q3W) schedule. Pomalidomide will be administered daily on Days 1 to 21 of each 28-day cycle, with dexamethasone administered once weekly (Days 1, 8, 15, and 22). Participants in both arms will be treated until disease progression, death, unacceptable toxicity, withdrawal of consent, and lost to follow-up or end of study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Participants must be 18 or older, at the time of signing the informed consent. In Republic of Korea, participants must be over 19 years of age inclusive, at the time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Histologically or cytologically confirmed diagnosis of Multiple myeloma (MM) as defined according to IMWG, and : Has undergone autologous stem cell transplant (SCT), or is considered transplant ineligible; Has received at least 2 prior lines of anti-myeloma treatments, including at least 2 consecutive cycles of both lenalidomide and a proteasome inhibitor (given separately or in combination), and must have documented disease progression on, or within 60 days of, completion of the last treatment or must be non-responsive while on last treatment, where non-responsive is defined as not achieving at least Minimal Response (MR) after 2 complete treatment cycles. In such cases lack of achieving of at least MR must be determined no earlier than at least 4 weeks after the last treatment.
* Has measurable disease with at least one of the following: Serum M-protein >=0.5 gram per deciliter (g/dL) (>=5 gram per Liter); Urine M-protein >=200 mg/24 hours; Serum free light chain (FLC) assay: Involved FLC level >=10 milligram per deciliter (mg/dL) (>=100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with a history of autologous SCT are eligible for study participation provided the following eligibility criteria are met: Transplant was >100 days prior to initiating study treatment; No active infection(s).
* Adequate organ system functions as defined: Absolute neutrophil count (ANC) >=1.0*10^9/L; Hemoglobin >= 8.0 g/dL; Platelets >= 50x10^9/L; Total bilirubin <=1.5* Upper limit of normal (ULN) (isolated bilirubin >1.5*ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent); ALT <=2.5*ULN; Estimated glomerular filtration rate (eGFR) >=30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2); Spot urine (albumin/creatinine ratios) <=500 milligram per gram (mg/g) (56 milligram per millimoles [mg/mmol]).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following during the intervention period and until 6 months after the last dose of study intervention to allow for clearance of any altered sperm: Refrain from donating sperm PLUS, either: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below depending on whether they are randomised to Arm 1 (belantamab mafodotin) or Arm 2 (pom/dex), even if they have undergone a successful vasectomy: Agree to use a male condom throughout study treatment including the 6 month follow-up period even if they have undergone a successful vasectomy and a female partner to use an additional highly effective contraceptive method with a failure rate of <1 percent per year when having sexual intercourse with a pregnant woman or a woman of childbearing potential who is not currently pregnant. Four weeks for male participants on Treatment Arm 2 (pom/dex).
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and agrees to abide by the following: Arm 1 (belantamab mafodotin): Use a contraceptive method that is highly effective (with a failure rate of <1 percent per year) which includes abstinence, preferably with low user dependency during the intervention period and for 4 months after the last dose of study treatment. Arm 2 (pom/dex): Due to pomalidomide being a thalidomide analogue with risk for embryofetal toxicity and prescribed under a pregnancy prevention/controlled distribution program, WOCBP participants will be eligible if they commit either to abstain continuously from heterosexual sexual intercourse or to use two methods of reliable birth control (one method that is highly effective), beginning 4 weeks prior to initiating treatment with pomalidomide, during therapy, during dose interruptions and continuing for at least 4 weeks following discontinuation of pomalidomide treatment. Two negative pregnancy tests must be obtained prior to initiating therapy. The first test should be performed within 10-14 days and the second test within 24 hours prior to prescribing pomalidomide therapy. And agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should confirm the effectiveness of the contraceptive method(s) ahead of the first dose of study intervention.
* All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events [NCI-CTCAE], version 5.0, 2017) must be <=Grade 1 at the time of enrollment, except for alopecia and Grade 2 peripheral neuropathy.

Exclusion Criteria:

* Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes); active plasma cell leukemia at the time of screening.
* Systemic anti-myeloma therapy or use of an investigational drug within <14 days or 5 half-lives, whichever is shorter, before the first dose of study intervention.
* Prior treatment with an anti-MM monoclonal antibody within 30 days prior to receiving the first dose of study intervention.
* Prior B cell maturation antigen (BCMA)-targeted therapy or prior pomalidomide treatment.
* Plasmapheresis within 7 days prior to the first dose of study intervention.
* Prior allogeneic stem cell transplant. (Participants who have undergone syngeneic transplant will be allowed only if no history of, or currently active, Graft-Versus-Host Disease [GvHD]).
* Any major surgery within the last 4 weeks.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil criteria as described in inclusion criteria.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance with study procedures.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Evidence of active mucosal or internal bleeding.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. (Stable chronic liver disease [including Gilbert's syndrome or asymptomatic gallstones] or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria)
* Participants with previous or concurrent malignancies other than multiple myeloma are excluded, unless the second malignancy has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease. (Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction).
* Evidence of cardiovascular risk including any of the following: Evidence of current clinically significant uncontrolled arrhythmias including clinically significant electrocardiogram (ECG) abnormalities including 2nd degree (Mobitz Type II) or 3rd degree atrioventricular block; History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening; Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; Uncontrolled hypertension.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin, pomalidomide, dexamethasone or any of the components of the study intervention.
* Pregnant or lactating female.
* Active infection requiring treatment.
* Known human immunodeficiency virus (HIV), unless the participant can meet all of the following criteria: Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL; CD4+ T-cell (CD4+) counts ≥350 cells/uL; No history of AIDS-defining opportunistic infections within the last 12 months.(Consideration must be given to ART and prophylactic antimicrobials that may have a drug-drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant)
* Participants with Hepatitis B will be excluded unless the following criteria can be met: If the participant is hepatitis B core antibody (HbcAb) positive or hepatitis B surface antigen (HbsAg) negative, then hepatitis B virus (HBV) deoxyribonucleic acid (DNA) should be undectectable at the time of screening; If HbsAg+ at screening or <=3 months prior to first dose of study treatment, then HBV DNA should be undetectable, highly effective antiviral treatment should be started ≥4 weeks prior to first dose of study treatment, exclusion of participants with cirrhosis and participants in Japan must test hepatitis B e antigen (HBeAg) and hepatitis B e antibody (HBeAb ).
* Positive hepatitis C antibody test result or positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria: Hepatitis C RNA test negative at Screening and successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period of at least 4 weeks (Hepatitis RNA is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing).
* Participants unable to tolerate thromboembolic prophylaxis.
* Current corneal epithelial disease except for mild punctate keratopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2027-03-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (86):
- United States (10):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Clifton Park, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (5):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Yvoir
- Brazil (6):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- GSK Investigational Site, Sofia, Bulgaria
- GSK Investigational Site, Edmonton, Alberta, Canada
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Xuzhou
  - GSK Investigational Site, Zhengzhou
- France (3):
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Poitiers
- Germany (2):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Tübingen
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari - Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Nyíregyháza
- Italy (9):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Catanzaro
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Ravenna
  - GSK Investigational Site, Roma
  - GSK Investigational Site, San Giovanni Rotondo FG
  - GSK Investigational Site, Siena
- Japan (11):
  - GSK Investigational Site, Shibuya-Ku, Tokyo
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Amersfoort, Netherlands
- GSK Investigational Site, Gdansk, Poland
- GSK Investigational Site, Kaluga, Russia
- South Korea (5):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (2):
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimopoulos MA, Hungria VTM, Radinoff A, Delimpasi S, Mikala G, Masszi T, Li J, Capra M, Maiolino A, Pappa V, Chraniuk D, Osipov I, Leleu X, Low M, Matsumoto M, Sule N, Li M, McKeown A, He W, Bright S, Currie B, Perera S, Boyle J, Roy-Ghanta S, Opalinska J, Weisel K. Efficacy and safety of single-agent belantamab mafodotin versus pomalidomide plus low-dose dexamethasone in patients with relapsed or refractory multiple myeloma (DREAMM-3): a phase 3, open-label, randomised study. Lancet Haematol. 2023 Oct;10(10):e801-e812. doi: 10.1016/S2352-3026(23)00243-0. PMID 37793771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on the primary analysis (and includes data up to a maximum of 27 months). Data collection is still ongoing and additional results will be provided after study completion.
Groups:
- Belantamab Mafodotin: Participants with relapsed/refractory multiple myeloma (RRMM) received at least 30 minutes intravenous infusion of 2.5 milligram/kilogram (mg/kg) belantamab mafodotin on day 1 of each 21-day cycle up to approximately 23 months.
- Pomalidomide Plus Dexamethasone: Participants with RRMM received 4 mg pomalidomide capsule daily on Days 1 to 21 of each 28-day cycle, along with 40 mg or at lower 20 mg (for participants >75 years of age) dose of dexamethasone tablet once weekly (Days 1, 8, 15 and 22) up to approximately 24 months.
Period: Overall Study
Arm/Group | Belantamab Mafodotin | Pomalidomide Plus Dexamethasone
Started (Intent-to Treat (ITT) population included all randomized participants whether or not randomized treatment was administered.) | 218 | 107
Safety Population (All randomized participants who took at least 1 dose of study intervention.) | 217 | 102
Completed | 84 | 38
Not Completed | 134 | 69
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Ongoing | 113 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin | Pomalidomide Plus Dexamethasone | Total
Number analyzed (Participants) | 218 | 107 | 325
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 66.3 (9.67) | 66.6 (9.68) | 66.4 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 41 | 141
  Male | 118 | 66 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 47 | 19 | 66
  Black Or African American | 3 | 1 | 4
  White | 162 | 84 | 246
  Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Investigator-assessed Response as Per International Myeloma Working Group (IMWG)
Description: PFS is time from randomization until earliest date of progressive disease (PD), or death due to any cause per investigator-assessed response per IMWG. PD is ≥25% increase from nadir in any of following: serum M-protein (absolute increase ≥0.5 gram per deciliter [g/dL]),urine M-protein(absolute increase ≥200 mg/24hr),difference between involved/uninvolved FLC levels (absolute increase >10 mg/dL) in patients without measurable serum and urine M-protein levels, or bone marrow plasma-cell percentage irrespective of baseline status (absolute increase ≥10%) in patients without measurable serum and urine M-protein levels and without measurable involved FLC levels; appearance of new lesion,≥50% increase in longest diameter of a lesion previously measured >1cm in short axis, or ≥50% increase from nadir in sum of products of two longest perpendicular diameters of more than 1 lesion; ≥50% increase in circulating plasma cells (minimum of 200 cells/microliter) if this is only measure of disease.
Time Frame: Up to 27 months
Population: Intent-to-treat population included all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 218 | 107
Months | 11.2 [6.4 to 14.5] | 7.0 [4.6 to 10.6]
Statistical Analysis 1: Comparison: Belantamab Mafodotin vs Pomalidomide Plus Dexamethasone; Test type: Other; p = 0.558, Log Rank; One-sided p-value from stratified log-rank test were adjusted for previous treatment with anti-CD38, ISS staging and number of prior lines of therapy; Stratified Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.72 to 1.47] — HR was estimated using the Cox Proportional Hazards. HR stratified log-rank test were adjusted for previous treatment with anti-CD38, international staging system (ISS) staging and number of prior lines of therapy

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death due to any cause.
Time Frame: 60 months
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed partial response (PR) or better per IMWG.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with a confirmed minimal response (MR) or better per IMWG.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from first documented evidence of PR or better until progressive disease (PD) per IMWG or death due to PD among participants who achieve confirmed PR or better.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time between the date of randomization and the first documented evidence of response (PR or better) among participants who achieve confirmed PR or better.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization until the earliest date of documented PD (per IMWG Response Criteria) or death due to PD.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Change From Baseline in Hematology Parameters: Absolute White Blood Cell Count (WBC), Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, and Neutrophils (Giga Cells Per Liter)
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Change From Baseline in Hematology Parameters: Red Blood Cell (RBC) Count and Reticulocyte Count (Trillion Cells Per Liter)
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Grams Per Liter)
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit (Proportion of Red Blood Cells in Blood)
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscular Volume (MCV) [Femtoliter]
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscular Hemoglobin (MCH) [Picograms]
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase (CK), Gamma Glutamyl Transferase (GGT), and Lactate Dehydrogenase (LDH)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters like ALT, AST, ALP, CK, GGT, and LDH [International units per Liter
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Calcium, Chloride, Glucose, Potassium, Sodium, Magnesium, Blood Urea Nitrogen (BUN), and Phosphorous (Millimoles Per Liter)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

17. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatinine, Direct Bilirubin, Total Bilirubin, Uric Acid (Micromoles Per Liter)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

18. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Total Protein (Grams Per Liter)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

19. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Specific Gravity (Ratio)
Description: Urine samples will be collected for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

20. Secondary Outcome: Change From Baseline in Urinalysis Parameters- Urine Potential of Hydrogen (pH) (Points on a Scale)
Description: Urine samples will be collected for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

21. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Glucose (Millimole Per Liter)
Description: Urine samples will be collected for the assessment of urinary glucose.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

22. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Protein (Grams Per Liter)
Description: Urine samples will be collected for the assessment of urinary protein.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

23. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Ketones (Millimoles Per Liter)
Description: Urine samples will be collected for the assessment of urinary ketones.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

24. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Blood (10^9 Cells Per Liter)
Description: Urine samples will be collected for the assessment of urinary blood.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

25. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Creatinine/Albumin Ratio (Ratio)
Description: Urine samples will be collected for the assessment of urinary creatinine/albumin ratio.
Time Frame: Baseline and up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

26. Secondary Outcome: Number of Participants With Abnormal Ocular Findings
Description: Participants will be assessed for any abnormal ocular findings.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

27. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin
Description: Blood samples will be collected for the analysis.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

28. Secondary Outcome: Plasma Concentrations of Total Monoclonal Antibody (mAb)
Description: Blood samples will be collected for the analysis.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

29. Secondary Outcome: Plasma Concentrations of Cys-mc Microtubular Inhibitor Monomethyl Auristatin-F (MMAF)
Description: Blood samples will be collected for the analysis.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

30. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADAs) Against Belantamab Mafodotin
Description: Blood samples will be collected for the analysis.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

31. Secondary Outcome: Titer of ADAs Against Belantamab Mafodotin
Description: Blood samples will be collected for the analysis.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

32. Secondary Outcome: Number of Participants With Symptomatic Adverse Effects Measured by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

33. Secondary Outcome: Number of Participants With Symptomatic Adverse Effects Measured by Ocular Surface Disease Index (OSDI)
Description: OSDI is a 12-item questionnaire designed to assesses both the frequency of dry eye symptoms and their impact on vision-related functioning. It is graded on a scale of 0-4, with 0 indicating none of the time, 1 for some of the time, 2 for half of the time, 3 for most of the time and 4 indicating all the time. A higher score represents greater symptoms severity.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

34. Secondary Outcome: European Organization for Research and Treatment of Cancer IL52 (EORTC IL52) Score
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems. A high score represents a high/healthy level of functioning.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

35. Secondary Outcome: Rate of Minimal Residual Disease (MRD)
Description: MRD negativity rate, defined as; the percentage of participants who are MRD negative by Next generation sequencing (NGS) method.
Time Frame: Up to 55 months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to 27 months. Data collection is still ongoing and additional results will be provided after study completion.
Description: All cause mortality, SAEs and non-serious adverse events were reported for the safety population that included all randomized participants who received at least 1 dose of any study intervention.
Arm/Group | Belantamab Mafodotin | Pomalidomide Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 83/217 | 38/102
Serious Adverse Events (participants affected / at risk) | 94/217 | 40/102
Other Adverse Events (participants affected / at risk) | 200/217 | 88/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin (N=217) | Pomalidomide Plus Dexamethasone (N=102)
Pneumonia (Infections and infestations) | 6 (6) | 8 (10)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary nocardiosis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 3 (3) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hyperammonaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (9) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Device extrusion (Product Issues) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin (N=217) | Pomalidomide Plus Dexamethasone (N=102)
Thrombocytopenia (Blood and lymphatic system disorders) | 70 (98) | 31 (61)
Anaemia (Blood and lymphatic system disorders) | 61 (78) | 30 (37)
Neutropenia (Blood and lymphatic system disorders) | 24 (47) | 39 (86)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 9 (19)
Lymphopenia (Blood and lymphatic system disorders) | 5 (8) | 7 (24)
Vision blurred (Eye disorders) | 86 (172) | 2 (2)
Dry eye (Eye disorders) | 61 (116) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 57 (129) | 2 (2)
Eye irritation (Eye disorders) | 50 (87) | 1 (2)
Photophobia (Eye disorders) | 46 (64) | 1 (1)
Visual acuity reduced (Eye disorders) | 41 (97) | 1 (1)
Eye pain (Eye disorders) | 35 (54) | 0 (0)
Keratopathy (Eye disorders) | 26 (29) | 1 (1)
Punctate keratitis (Eye disorders) | 23 (44) | 0 (0)
Visual impairment (Eye disorders) | 13 (25) | 0 (0)
Cataract (Eye disorders) | 12 (14) | 5 (6)
Keratitis (Eye disorders) | 12 (14) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 33 (37) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 30 (32) | 5 (8)
Platelet count decreased (Investigations) | 27 (32) | 12 (19)
Gamma-glutamyltransferase increased (Investigations) | 22 (24) | 5 (6)
Neutrophil count decreased (Investigations) | 17 (35) | 14 (34)
Alanine aminotransferase increased (Investigations) | 14 (16) | 8 (17)
White blood cell count decreased (Investigations) | 12 (19) | 9 (21)
Blood creatinine increased (Investigations) | 10 (11) | 6 (7)
Lymphocyte count decreased (Investigations) | 8 (15) | 6 (9)
Pyrexia (General disorders) | 34 (47) | 9 (11)
Fatigue (General disorders) | 18 (19) | 15 (15)
Chills (General disorders) | 13 (16) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 10 (12)
Nausea (Gastrointestinal disorders) | 25 (32) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 22 (27) | 11 (14)
Vomiting (Gastrointestinal disorders) | 16 (22) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (12) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 10 (11)
COVID-19 (Infections and infestations) | 24 (24) | 9 (9)
Urinary tract infection (Infections and infestations) | 12 (17) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (16) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 15 (25) | 0 (0)
Hypertension (Vascular disorders) | 13 (13) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 11 (14) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04162210/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04162210/SAP_001.pdf